CLINICAL TRIAL: NCT04748341
Title: The Efficacy of Pedagogical Framework (Learn, See, Practice, Prove, Do, Maintain) on Knowledge, Skill, and Self-Efficacy of Nursing Students Regarding Neonatal Resuscitation.
Brief Title: The Impact of Pedagogical Framework in Education of Neonatal Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Mishal Liaqat, Principal Investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-UOL-FAHS/775/2020
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Nursing Students Education on Neonatal Resuscitation
MeSH Terms: interventions — Educational Status; Vision, Ocular; Benzocaine

STUDY DESIGN:
Intervention Model Description: The study design is a Single-blind randomized control trial conducted in the College of Nursing, Allama Iqbal Medical College, Lahore, Pakistan. A sample size of 72 nursing students (36 in each group) will be taken through simple random sampling. The students allocated from each professional in group A and group B through the Lottery method. Allocation of participants was concealed using envelop method. A total of 6 weeks of intervention will be provided to both groups. Group A will be taught through the two steps traditional method (2 lectures/week + 1 skill lab/week). On the contrary Group B will learn through the 6-step method constituted 2 lecture/week + video + 2skill lab/week (1 session under instructor + 1 session for skill maintenance).
Who Masked: Outcomes Assessor
Masking Description: The data will be collected at two points in time. 1st-time data will be collected as a pre-test before the educational intervention. The 2nd-time data will be collected after 6 weeks of educational intervention. Two facilitator evaluators will be trained regarding the scoring of each scale in a two-hour workshop before data collection. All the students were allotted code after allocation. Only the principal investigator knows the allocation status of each student code. The skill was tested through simulation scenarios in the skill lab. The facilitators, who assessed the student's skills, endure uninformed regarding the student's allocation status and sequence of the scenario in the pre-and post-data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Group (Active Comparator): Group A will be taught through the two steps traditional method (2 lectures/week + 1 skill lab/week). First, learn through didactic Lectures and then practice skills on the Mannequins. The educational lecture content will be the same for both groups.
  Interventions: Other: Traditional Method
- Pedagogical Group (Experimental): Group B will learn through the 5-step method [ 2 lectures/week + video + 2skill lab/week (1 session under instructor + 1 session for skill maintenance)], learn skill, see the video on resuscitation, practice on simulator, prove through practice, observe skill on clinical rotation and lastly maintain it through clinical supplemented with simulation.
  Interventions: Other: Pedagogical Framework (Learn, See, Practice, Prove, Do, and Maintain)

INTERVENTIONS:
Other: Pedagogical Framework (Learn, See, Practice, Prove, Do, and Maintain) — The "Learn, See, Practice, Prove, Do, and Maintain" (LSPPDM) pedagogy is acting as a guiding path for educators in teaching and learning procedural skills. It is synthesized after intensely reviewing the literature comprises steps. In the 1st step, learners learn through didactic lectures, further proceeding to see procedural videos. The 3rd step, "Practice" expose learners to perform the skill on a simulator. In the 4th step "Prove" the learner proves the skill. The 5th step Do comprise real-life exposure through the clinical rotation. Then, finally the 6th step"Maintain" the learner maintains skill supplemented with simulation as needed.
  Arms: Pedagogical Group
Other: Traditional Method — The traditional method group learns through 2-step method.
  1. didactic lectures on neonatal resuscitation were delivered.
  2. Practice skill on mannequins
  Arms: Traditional Group

SUMMARY:
Virtually 10% of newborns suffer respiratory distress at birth thus need intervention from proficient health professionals. Pakistan is one of the top ten countries that carry two-thirds of the global burden of neonatal deaths. It is suggested that most of these deaths can be prevented through the provision of trained emergency birth attendants, in which education plays an integral role. Since its inception in the neonatal resuscitation program, we are still in the struggle to find out the best strategies to disseminate NRP knowledge, training, and guidelines that promise the best outcome. Hence, little published data on this phenomenon is available regarding undergraduate students. That determines the best way to educate them in performing the skills that urgently require an infrequent needed such as neonatal resuscitation. Therefore, this study intended to address this gap in the education of neonatal resuscitation through two different approaches. One is a traditional 2-step method and the other is an adapted Pedagogical framework (Lean, See, Practice, Prove, Do and Maintain).

DETAILED DESCRIPTION:
Globally, nurses are the largest workforce in the healthcare system that are directly engaged in the provision of newborn care. They should be conversant and competent in neonatal resuscitation. However, the majority of nurses are not skillful in the respective field. The situation is not very different when we are talking about nursing students. Who are our future workforce, hence are found incompetent in emergency newborn management and neonatal resuscitation. It is well documented that effective educational programs in preservice settings such as schools of midwifery, nursing, and medicine, established more active forms of lifelong learning to improve the quality of care. While the transformation of theoretical knowledge into clinical practice requires effective teaching in the field of resuscitation is a vital element for all undergraduate students. However, like many other developing countries in Pakistan, mostly traditional methods are following in nursing education. While the traditional method of teaching is insufficient to meet the educational demands of nursing students in clinical practice. Hence, Nursing students often are unprepared and lacking confidence in simple, yet life-saving procedures such as neonatal resuscitation. Therefore, incorporating an effective model and framework in nursing education is needed that could enhance nursing students' skills and improve clinical outcomes. The "Learn, See, Practice, Prove, Do, and Maintain" (LSPPDM) pedagogy is one of such frameworks synthesized after intensely reviewing the literature. This framework is acting as a guiding path for educators in teaching and learning procedural skills. As Knowledge is considering a prerequisite for competence in skill performance and to evaluate the effectiveness of an educational program self -efficacy measurement is an important tool. Thus, the important variables knowledge, self-efficacy, and skill have been selected for this study. Thus, the study objective will be:

To compare the knowledge, skill, and self-efficacy among undergraduate nursing students learning of neonatal resuscitation through "Learn, See, Practice, Prove, Do, Maintain pedagogy" as compared to those who will learn through the traditional method.

This study will contribute essentially to determine the effectiveness of an adapted pedagogical framework in the teaching and learning of neonatal resuscitation skills, especially in a resource-limited society. Moreover, the study findings will help the organization to develop strategies for improving nursing education.

ELIGIBILITY:
Inclusion Criteria:

* Are currently enrolled in the Bachelor of Science in Nursing (4 years) 3rd and 4th Professional.
* Those willing to attend the full course of neonatal resuscitation.
* Having age 18-25 years.
* Those willing to give informed consent.

Exclusion Criteria:

* Will be on leave from that period
* Have already received any educational training on neonatal resuscitation.
* Working as Nursing Assistants in Clinical Setting.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mishal Liaqat, Principal Investigator — Lahore School of Nursing, The University of Lahore; Muhammad Hussain, Study Chair — Lahore School of Nursing, The University of Lahore; Muhammad Afzal, Study Chair — Lahore School of Nursing, The University of Lahore; Amir Gillani, Study Director — Faculty of Allied Health Sciences, The University of Lahore
Locations (1):
- College of Nursing, Allama Iqbal Medical College., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liaqat M, Hussain M, Afzal M, Altaf M, Khan S, Gilani SA, Liaqat I. Efficacy of pedagogical framework in neonatal resuscitation skill learning in a resource-limited setting: a randomized controlled trial. BMC Med Educ. 2021 Aug 18;21(1):436. doi: 10.1186/s12909-021-02846-x. PMID 34407810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: initially, 62 participants (31 in each group) were recruited. one participant from each group was lost in follow-up due to some personal reasons. The final sample size remained 60 (30 in each group).
Pre-assignment Details: Two participants were dropped in the follow-up for personal reasons one was not attending the full course of intervention and the other was absent on the days of evaluation. Thus, yielding a total of 60 participants (30 in each group).
Groups:
- Traditional Group: Group A will be taught through the two steps traditional method (2 lectures/week + 1 skill lab/week). First, learn through didactic Lectures and then practice skills on the Mannequins. The educational lecture content will be the same for both groups.
  Traditional Method: The traditional method group learns through 2-step method.
  1. didactic lectures on neonatal resuscitation were delivered.
  2. Practice skill on mannequins
- Pedagogical Group: Group B will learn through the 6-step method [ 2 lectures/week + video + 2skill lab/week (1 session under instructor + 1 session for skill maintenance)], learn skill, see the video on resuscitation, practice on simulator, prove through practice, observe skill on clinical rotation and lastly maintain it through clinical supplemented with simulation.
  Pedagogical Framework (Learn, See, Practice, Prove, Do, and Maintain): The "Learn, See, Practice, Prove, Do, and Maintain" (LSPPDM) pedagogy is acting as a guiding path for educators in teaching and learning procedural skills. It is synthesized after intensely reviewing the literature comprises steps. In the 1st step, learners learn through didactic lectures, further proceeding to see procedural videos. The 3rd step, "Practice" expose learners to perform the skill on a simulator. In the 4th step "Prove" the learner proves the skill. The 5th step Do comprise real-life exposure through the clinical rotation. Then, finally the 6th step"Maintain" the learner maintains skill supplemented with simulation as needed.
Period: Overall Study
Arm/Group | Traditional Group | Pedagogical Group
Started | 31 | 31
Completed | 30 | 30
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Group | Pedagogical Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (0.75) | 21.9 (1.1) | 22 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Year of Professional Education [Number; unit: participants] — The Year of professional education describes that how many students were in the 3rd year and 4th year in both traditional and pedagogy groups. It will describe the number of participants studied in the 3rd year and the number of participants studied in the 4th year.
  participants
    3rd year | 14 | 15 | 30
    4th year | 16 | 15 | 30
Primary Language [Number; unit: participants]
  Urdu | 29 | 29 | 58
  Punjabi | 1 | 1 | 2
Marital Status [Number; unit: participants]
  Unmarried | 29 | 30 | 59
  Married | 1 | 0 | 1
Residential Area [Number; unit: participants]
  Rural | 3 | 2 | 5
  Urban | 27 | 28 | 55
Division in previous results [Number; unit: participants] — Division in previous results means that the number of participants who got 1st division (> 60% marks) in the previous year exams and the number of participants who got 2nd division (< 60% marks) in the previous year exam.
  participants
    First | 28 | 30 | 58
    Second | 2 | 0 | 2
Previous neonatal resuscitation exposure [Number; unit: participants] — Previous neonatal resuscitation exposure means the number of participants who had seen neonatal resuscitation previously during their clinical rotation.
  participants
    Yes | 5 | 3 | 8
    No | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Questionnaire
Description: knowledge is considering awareness of Neonatal resuscitation. It will be measured through a 17-item multiple-choice question adopted from Knowledge Question total score ranged from 0 to 17. A higher score means have more knowledge.
Time Frame: before intervention and 6 weeks after intervention
Population: All participants were randomly assigned to traditional and pedagogy groups. The analysis was done before and 6 weeks after the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Group | Pedagogical Group
Number analyzed (Participants) | 30 | 30
score on a scale
  before 6 weeks (pre data) | 5.90 (1.95) | 5.87 (1.87)
  After 6 weeks (Post data) | 9.97 (1.22) | 13.33 (1.30)

2. Primary Outcome: Self-efficacy for Neonatal Resuscitation (SENR)
Description: The SENR instrument is a 23-item scale that measured nursing students' perception of confidence in their capabilities in neonatal resuscitation. All SENR items were valued on a 10-point Likert scale. The total score ranged from 0 to 230. A higher score means have more self-efficacy.
Time Frame: before intervention and 6 weeks after intervention
Population: Participants were randomly assigned into traditional and pedagogy group and were analyzed two times before and 6 weeks after the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Group | Pedagogical Group
Number analyzed (Participants) | 30 | 30
score on a scale
  Before 6 weeks (pre data) | 96.1 (35.5) | 95.9 (37.6)
  After 6 weeks (Post data) | 186.6 (25.3) | 188.6 (24.2)

3. Primary Outcome: Neonatal Resuscitation Checklist
Description: A 30 items checklist will be used. Each of the correct actions was graded as 1=yes and for wrong action 0=no. The total score ranged from 0 to 30. The total score ranged from 0 to 30. A higher score means have more skill.
Time Frame: before intervention and 6 weeks after intervention
Population: Participants were randomly assign into traditional and pedagogy group and were assessed for skill before and 6 weeks after the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Group | Pedagogical Group
Number analyzed (Participants) | 30 | 30
score on a scale
  Before intervention (pre data) | 3.30 (1.18) | 3.37 (1.10)
  6 weeks after intervention (post data) | 16.20 (2.40) | 24.27 (3.47)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Traditional Group | Pedagogical Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT04748341/Prot_SAP_ICF_000.pdf